CLINICAL TRIAL: NCT04916743
Title: The Effect of Intradialytic Exercise on Calcium, Phosphorus and Parathyroid Hormone: A Randomized Controlled Trial
Brief Title: The Effect of Exercise on Blood Parameters Related to Dialysis Patients' Survival
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA21HD-2-04
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Diseases; End Stage Renal Disease; Hemodialysis
Keywords: Mortality; Mortality Rate; Survival; Cardiovascular Disease; Osteoporosis; Bone Mineral Disorders; Exercise during dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Cardiovascular Diseases; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way.
Who Masked: Outcomes Assessor
Masking Description: The lab tech will be blind to whether the sample under evaluation belongs to the intervention group or the control group. Outcome adjudicators, and data analysts will be kept blinded to the allocation. Moreover, all investigators, staff, and participants will be kept masked to outcome measurements and trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The patients will participate in intradialytic exercise 3 times a week for 24 weeks.
  Interventions: Other: Intradialytic exercise group
- Control group (No Intervention): The patients will receive regular care and treatment in every dialysis sessions without any intradialytic exercise.

INTERVENTIONS:
Other: Intradialytic exercise group — Participants will do concurrent exercise (a combination of aerobic exercise and resistance training) for 30-60 minutes during the second hour of their routine hemodialysis sessions. To determine the intensity of the prescribed exercise, maximum heart rate is used for aerobic workout and 5 Repetitions Maximum (5RM) for resistance protocols. Exercises will be performed at a moderate exercise intensity (12-14 on the Borg RPE Scale). All protocols are tailor-made based on each individual's needs and physical abilities.
  Arms: Exercise group

SUMMARY:
The purpose of this study is to check if patients' exercise during their dialysis sessions can improve the blood parameters which affect the heart disease and osteoporosis, so that we can help patients live longer.

DETAILED DESCRIPTION:
Dialysis patients suffer from a number of problems, one of which is reduced ability, decreased functional capacity, and consequently reduced physical capability. Forced inactivity due to immobility in dialysis sessions and the need to rest and relieve fatigue for a few hours after each session cause patients to become more inactive day by day, and according to various studies, inactivity in these patients along with reduced physical capabilities increase the risk of cardiovascular disease (CVD), which is a risk factor for mortality in these patients.

On the other hand, inactivity is an independent predictor of hospitalization and mortality in these patients.

The mortality rate of dialysis patients is much higher than that of healthy people, to the extent that it is reported to be about 10 to 30 times higher. The life expectancy of these patients is between 30 and 50 percent lower than that of people without the same age and sex. Dialysis patients suffer from many CVDs such as high blood pressure, vascular disease, congestive heart failure and arrhythmias. CVDs in patients are related to traditional risk factors such as diabetes, hypertension, sedentary lifestyle and non-traditional risk factors such as anemia, inflammation, abnormal calcium metabolism and phosphorus and oxidative stress. Studies have shown that high levels of calcium, phosphorus , calcium- phosphorus product and parathyroid hormone are associated with fatal and non-fatal cardiovascular events and all-cause mortality in dialysis patients.

One of the most common complications of chronic kidney disease is hypophosphatemia. Phosphate metabolism is regulated by the interaction of the kidneys, bones and intestines. This balance is impaired in kidney patients and the calcification process occurs through disturbances in the regulation of calcium, phosphate, and hyperparathyroidism. Hyperparathyroidism is considered as one of the aggravating causes of anemia as well as resistance to erythropoietin treatment in hemodialysis patients. Due to the effect of parathyroid hormone in the regulation of calcium and the anabolic and catabolic role of the bones, the regulation of this hormone is essential for all people, especially dialysis patients.

Human studies have shown that the regulation of parathyroid hormone and calcium and phosphorus metabolism are dependent on physical activity, and they have introduced exercise as an effective way to regulate this hormone. Considering the various effects of exercise on dialysis patients, a study has been designed to investigate the effect of concurrent exercise during dialysis on changes in calcium levels, phosphorus, calcium-phosphorus product, and parathyroid hormone.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis history ≥ 1 year
* Without myocardial infarction within past 3 months
* Regular dialysis 3 times a week
* Ability to consent
* Doctor's consent

Exclusion Criteria:

* Unstable cardiac status (angina, decompensated congestive heart failure, severe arteriovenous stenosis, uncontrolled arrhythmias, etc.)
* Active infection or acute medical illness
* Hemodynamic instability
* Labile glycemic control
* Unable to exercise (lower extremity amputation with no prosthesis)
* having severe musculoskeletal pain at rest or with minimal activity
* Unable to sit, stand or walk unassisted (walking device such as cane or walker allowed)
* Having shortness of breath at rest or with activities of daily living (NYHA Class IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Rate of changes of Calcium for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Phosphorus for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Parathyroid Hormones for 6 months | Pre_test and every 3 months for 6 months

SECONDARY OUTCOMES:
Rate of changes of Calcium-Phosphorous product for 6 months | Pre_test and every 3 months for 6 months
Rate of changes of Alkaline Phosphatase for 6 months | Pre_test and every 3 months for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Principal Investigator — Pardis Specialized Wellness Institute; Mohammad Ali Tabibi, Dr, Study Director — Pardis Specialized Wellness Institute; Shahrzad Amirian Farsani, Principal Investigator — Pardis Specialized Wellness Institute
Locations (2):
- Iran (2):
  - Abolfazl medical center, Isfahan
  - Pardis specialized wellness institute, Isfahan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the published article, after deidentification are to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: The IPD will be available only for our colleagues in Global Renal Exercise (GREX) as long as they have acceptable reasons for requiring the data.

REFERENCES:
- [Background] Parker K. Intradialytic Exercise is Medicine for Hemodialysis Patients. Curr Sports Med Rep. 2016 Jul-Aug;15(4):269-75. doi: 10.1249/JSR.0000000000000280. PMID 27399824
- [Background] K/DOQI Workgroup. K/DOQI clinical practice guidelines for cardiovascular disease in dialysis patients. Am J Kidney Dis. 2005 Apr;45(4 Suppl 3):S1-153. No abstract available. PMID 15806502
- [Background] Milam RH. Exercise Guidelines for Chronic Kidney Disease Patients. J Ren Nutr. 2016 Jul;26(4):e23-5. doi: 10.1053/j.jrn.2016.03.001. No abstract available. PMID 27318109
- [Background] Noordzij M, Korevaar JC, Boeschoten EW, Dekker FW, Bos WJ, Krediet RT; Netherlands Cooperative Study on the Adequacy of Dialysis (NECOSAD) Study Group. The Kidney Disease Outcomes Quality Initiative (K/DOQI) Guideline for Bone Metabolism and Disease in CKD: association with mortality in dialysis patients. Am J Kidney Dis. 2005 Nov;46(5):925-32. doi: 10.1053/j.ajkd.2005.08.013. PMID 16253734
- [Background] Pu J, Jiang Z, Wu W, Li L, Zhang L, Li Y, Liu Q, Ou S. Efficacy and safety of intradialytic exercise in haemodialysis patients: a systematic review and meta-analysis. BMJ Open. 2019 Jan 21;9(1):e020633. doi: 10.1136/bmjopen-2017-020633. PMID 30670499
- [Background] Noordzij M, Korevaar JC, Dekker FW, Boeschoten EW, Bos WJ, Krediet RT, Bossuyt PM, Geskus RB; NECOSAD study group. Mineral metabolism and mortality in dialysis patients: a reassessment of the K/DOQI guideline. Blood Purif. 2008;26(3):231-7. doi: 10.1159/000118847. Epub 2008 Feb 28. PMID 18305386
- [Background] Stevens LA, Djurdjev O, Cardew S, Cameron EC, Levin A. Calcium, phosphate, and parathyroid hormone levels in combination and as a function of dialysis duration predict mortality: evidence for the complexity of the association between mineral metabolism and outcomes. J Am Soc Nephrol. 2004 Mar;15(3):770-9. doi: 10.1097/01.asn.0000113243.24155.2f. PMID 14978180
- [Background] Bohm CJ, Ho J, Duhamel TA. Regular physical activity and exercise therapy in end-stage renal disease: how should we move forward? J Nephrol. 2010 May-Jun;23(3):235-43. PMID 20383863
- [Background] Aucella F, Gesuete A, Battaglia Y. A "nephrological" approach to physical activity. Kidney Blood Press Res. 2014;39(2-3):189-96. doi: 10.1159/000355796. Epub 2014 Jul 29. PMID 25118037
- [Background] Tuysuz ME, Dedemoglu M. Calcium phosphate product level as a predictor for arteriovenous fistula re-operations in patients with chronic renal failure. Vascular. 2019 Jun;27(3):284-290. doi: 10.1177/1708538118814611. Epub 2018 Nov 21. PMID 30463499
- [Background] Fernandez-Martin JL, Martinez-Camblor P, Dionisi MP, Floege J, Ketteler M, London G, Locatelli F, Gorriz JL, Rutkowski B, Ferreira A, Bos WJ, Covic A, Rodriguez-Garcia M, Sanchez JE, Rodriguez-Puyol D, Cannata-Andia JB; COSMOS group. Improvement of mineral and bone metabolism markers is associated with better survival in haemodialysis patients: the COSMOS study. Nephrol Dial Transplant. 2015 Sep;30(9):1542-51. doi: 10.1093/ndt/gfv099. Epub 2015 Apr 28. PMID 25920921
- [Background] Fujii H. Association between Parathyroid Hormone and Cardiovascular Disease. Ther Apher Dial. 2018 Jun;22(3):236-241. doi: 10.1111/1744-9987.12679. Epub 2018 Apr 30. PMID 29707916
- [Background] Tentori F, Blayney MJ, Albert JM, Gillespie BW, Kerr PG, Bommer J, Young EW, Akizawa T, Akiba T, Pisoni RL, Robinson BM, Port FK. Mortality risk for dialysis patients with different levels of serum calcium, phosphorus, and PTH: the Dialysis Outcomes and Practice Patterns Study (DOPPS). Am J Kidney Dis. 2008 Sep;52(3):519-30. doi: 10.1053/j.ajkd.2008.03.020. Epub 2008 Jun 2. PMID 18514987
- [Background] Kalantar-Zadeh K, Kuwae N, Regidor DL, Kovesdy CP, Kilpatrick RD, Shinaberger CS, McAllister CJ, Budoff MJ, Salusky IB, Kopple JD. Survival predictability of time-varying indicators of bone disease in maintenance hemodialysis patients. Kidney Int. 2006 Aug;70(4):771-80. doi: 10.1038/sj.ki.5001514. Epub 2006 Jul 5. PMID 16820797
- [Background] Block GA, Klassen PS, Lazarus JM, Ofsthun N, Lowrie EG, Chertow GM. Mineral metabolism, mortality, and morbidity in maintenance hemodialysis. J Am Soc Nephrol. 2004 Aug;15(8):2208-18. doi: 10.1097/01.ASN.0000133041.27682.A2. PMID 15284307
- [Background] Huang M, Lv A, Wang J, Xu N, Ma G, Zhai Z, Zhang B, Gao J, Ni C. Exercise Training and Outcomes in Hemodialysis Patients: Systematic Review and Meta-Analysis. Am J Nephrol. 2019;50(4):240-254. doi: 10.1159/000502447. Epub 2019 Aug 27. PMID 31454822
- [Background] Wilund K, Thompson S, Bennett PN. A Global Approach to Increasing Physical Activity and Exercise in Kidney Care: The International Society of Renal Nutrition and Metabolism Global Renal Exercise Group. J Ren Nutr. 2019 Nov;29(6):467-470. doi: 10.1053/j.jrn.2019.08.004. Epub 2019 Oct 4. No abstract available. PMID 31591041
- [Background] Lombardi G, Ziemann E, Banfi G, Corbetta S. Physical Activity-Dependent Regulation of Parathyroid Hormone and Calcium-Phosphorous Metabolism. Int J Mol Sci. 2020 Jul 29;21(15):5388. doi: 10.3390/ijms21155388. PMID 32751307
- [Derived] Tabibi MA, Wilund KR, Salimian N, Nikbakht S, Soleymany M, Roshanaeian Z, Nazemi F, Ahmadi S. The effect of intradialytic exercise on calcium, phosphorus and parathyroid hormone: a randomized controlled trial. BMC Nephrol. 2023 Sep 20;24(1):276. doi: 10.1186/s12882-023-03327-7. PMID 37730530